CLINICAL TRIAL: NCT06663202
Title: Fibre-Retention Osseous Resective Surgery (FibReORS) Vs Conservative Surgery with or Without Papilla Preservation Technique for the Treatment of Residual Pockets: a 5-year Randomized Clinical Trial
Brief Title: Osseous Resective Surgery Vs Conservative Surgery with or Without Papilla Preservation Technique
Acronym: FibReORS vs AF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Mario Aimetti, Associate Professor, University of Turin, Italy
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TurinPerioSurgery
Record Dates: First submitted 2024-10-22; First posted 2024-10-29 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Fiber Retention Osseous Resective Surgery (Experimental): Paramarginal incisions both on buccal and lingual/palatal sides with bone remodelling preserving the supracrestal fibers
  Interventions: Procedure: Fiber retention osseous resective surgery
- Papilla preservation flap (Active Comparator): Access flap for open flap debridement using intrasulcular incisions and papilla preservation approaches to preserve the entire interdental tissues
  Interventions: Procedure: Papilla preservation flap
- Conventional surgery (Active Comparator): Access flap for open flap debridement using a conventional modified Widman flap procedure
  Interventions: Procedure: Widman flap procedure

INTERVENTIONS:
Procedure: Fiber retention osseous resective surgery — At the buccal and lingual sides, paramarginal or intrasulcular incisions will be made based on probing pocket depth values and the width of keratinised tissues.
  Thinned palatal flap technique will be performed on the palatal side. Bone remodelling will be carefully made using manual or rotary instruments in order to reshape positive attached fibres/bony architecture utilising the FibReORS technique, great attention will be made to distinguish between inflammatory granulation tissue and connective tissue fibres attached to root cementum by means of periodontal probe. Flaps will be positioned at the level of the alveolar crest without tension.
  Arms: Fiber Retention Osseous Resective Surgery
Procedure: Papilla preservation flap — Surgical access will be obtained using modified papilla preservation techniques and when interproximal space is narrow (less than 3mm in width) incision will be made using the simplified papilla preservation flap. Both flaps buccal and lingual/palatal will be elevated in any case to allow root surface cleaning and defects debridement under direct vision. Minimally invasive flap elevation preventing to damage inter proximal tissues with the preservation of the papilla. Defects debridement with mini-curettes. Root surface debridement with ultrasonic debridement with periotip and mini-curettes. Flaps will be positioned at the pre-surgical level without any tension. Monofilament non-resorbable 5-0 e-PTFE suturing material will be used. Suturing will be performed with external vertical mattress sutures to achieve primary intention closure.
  Arms: Papilla preservation flap
Procedure: Widman flap procedure — Surgical access will be obtained using the modified Widman flap technique. Intrasulcular incision will be done on both buccal and lingual/palatal sides without attempting to preserve the interdental tissues and interdental tissues will be removed. Both flaps buccal and lingual/palatal will be elevated at full thickness in any case to allow root surface cleaning and defects debridement under direct vision, a vertical releasing incision could be made when needed.
  Defects debridement with mini-curettes. Root surface debridement with ultrasonic debridement with periotip and mini-curettes. Flaps will be positioned at the level of the alveolar crest without tension. Monofilament nonresorbable 5 - 0 e/PTFE suturing material will be used. Suturing will be performed with single interrupted sutures.
  Arms: Conventional surgery

SUMMARY:
The primary aim of the study is to evaluate the efficacy of either fibre retention osseous resective surgery (FibReORS) or conservative surgery with or without PPT in the treatment of deep residual pockets ≥ 6 mm in stage III-IV periodontitis patients after cause related therapy (step II) in terms of endpoints of therapy and other secondary outcomes at different time intervals (1, 3 and 5 years). Moreover, the study aims to evaluate the stability of the results obtained for the different surgical approaches over a 5 years follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of stage III/IV periodontitis.
* Completed steps I-II periodontal therapy at least 6 weeks before.
* Full Mouth Plaque Score less than 15% at re-evaluation.
* Full Mouth Bleeding Score less than 15% at re-evaluation.
* Posterior sextant with residual PPD ≥ 6 mm at ≥ 2 natural teeth (third molars excluded).
* Signed informed consent.

Exclusion Criteria:

* Compromised general health which contraindicates the study procedures (ASA III-VI patients).
* Systemic diseases/medications which could influence the outcome of the therapy (e.g. uncontrolled diabetes mellitus, non-plaque-induced gingival diseases, antiepileptic drugs (phenytoin and sodium valproate), certain calcium channel-blocking drugs (e.g., nifedipine, verapamil, diltiazem, amlodipine, felodipine), immunoregulating drugs (e.g., ciclosporine), and high-dose oral contraceptives).
* Pregnant or nursing women.
* Presence of tooth mobility ≥ class 2.
* Presence of furcation involvement ≥ II degree (Hamp 1975) at the affected teeth.
* Presence of deep infrabony defects (≥ 3 mm) at the involved sextant.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-11-15 (Estimated); Primary Completion 2030-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Pocket closure | 5 years
  Defined as probing pocket depth (PPD) of 3 mm or less or PPD of 4 mm with the absence of Bleeding on Probing in sites with PPD equal or more than 6 mm at baseline.

SECONDARY OUTCOMES:
Mean Probing Pocket Depth changes | 5 Years
  Defined as the mean changes in Probing pocket depth (distance in mm from the gingival margin to the bottom of the probable sulcus) at the involved sextant with respect to baseline.
Mean Clinical Attachment Level changes | 5 years
  Defined as the mean changes in Clinical Attachment Level (distance in mm from the Cemento Enamel Junction to the bottom of the probable sulcus) at the involved sextant with respect to baseline.
Mean recession changes | 5 years
  Defined as the changes in recession (distance in mm from cemento enamel junction to the gingival margin).
Tooth Retention | 5 years
  Number of teeth in the treated sextant present at the last follow-up evaluation.
Number of instrumentation re-intervention | 5 years
  Number of re-instrumentation interventions during supportive periodontal therapy performed at sites with incomplete outcome.

OTHER OUTCOMES:
Pain after surgery | 14 days
  The patient will self report pain on a 10 cm visual analog scale [0-100].
Discomfort during surgery | Immediately after surgery.
  Self reported on a 10 cm visual analog scale [0-100].